CLINICAL TRIAL: NCT00013819
Title: Exposure, Dose, Body Burden and Health Effects of Lead
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 7198-CP-001
Record Dates: First submitted 2001-03-29; First posted 2001-03-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Lead Poisoning
Keywords: lead poisoning; central nervous system; peripheral nervous system; occupational health; genetic susceptibility
MeSH Terms: conditions — Lead Poisoning; Genetic Predisposition to Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a study of the effects that lead has on the health of the central nervous system (for example, memory), peripheral nervous system (for example, sensation and strength in the hands and fingers), kidneys, blood pressure, and the blood forming system. A total of 803 lead workers and 135 persons without occupational lead exposure are being studied in South Korea. Lead in the body is being assessed by measurement of blood lead, chelatable lead (an estimate of lead in the tissues), and lead in bone. Subjects are tested three times each over three years. Several genetic factors are also being assessed for the role they play in the health effects of lead. These genes are known to differ among individuals. We are interested to know whether different forms of the same genes can modify the effect lead has on health.

ELIGIBILITY:
Lead workers in South Korea in one of 26 specific lead-using facilities.

Population controls in South Korea.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 944
Dates: Start 1997-02; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)